CLINICAL TRIAL: NCT03984162
Title: Influence of Individualized, Spiroergometry Guided, Structural Training on Cardiopulmonary Exercise Capacity in Patients With a Left Ventricular Assist Device
Brief Title: Influence of Individualized Training on Cardiopulmonary Exercise Capacity in LVAD Patients
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ_KA_016_LKW
Record Dates: First submitted 2019-03-11; First posted 2019-06-12 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the influence of an individualized, spiroergometry- guided training on cardiopulmonary fitness in patients with a left ventricular assist device (LVAD). Secondary endpoints are to establish an individualized but standardized and clinically safe training protocol for patients with LVAD implanted. The investigators aim to include sixty patients with first implanted LVAD to be included in this study over a term of 24 months. All study participants will perform cardiopulmonary exercise testing (CPET) at baseline before randomization and at the end of the study. Randomization into a control group and a training group will be performed subsequently. The control group will receive standard physiotherapeutic treatment as usual, including respiratory supportive therapy, mobilization, stability and coordination training. The training group will additionally receive five individualized training sessions on ergometer per week. Three sessions will consist of interval training; the other two sessions will consist of endurance training. The training group will further perform CPET every two weeks in order to adjust their individual training protocol.

DETAILED DESCRIPTION:
b.) Current European guidelines for prevention of cardiovascular disease recommend regular training for patients suffering from any cardiovascular disease. Studies have shown that regular training results in an improvement of cardiopulmonary exercise capacity. Objective parameters such as peak VO2 and VE/ VCO2 slope can be positively influenced by training in patients with heart failure. Only few studies suggest a beneficial impact on exercise capacity in patients with an implanted ventricular assist device (LVAD), but literature on this topic is scarce. So far there are no recommendations for a standardized exercise protocol for LVAD.

The aim of this prospective monocentric study is to examine the influence of an individualized, spiroergometry- guided training protocol on cardiopulmonary fitness in patients with an implanted LVAD. Secondary endpoints are to establish an individualized but standardized and clinically safe training protocol for patients with implanted LVAD.

The investigators goal is to include sixty patients with first implanted LVAD in this study over a term of 24 months. After providing written informed consent, randomization into a control group and into a training group will be conducted. All study participants will perform cardiopulmonary exercise testing (CPET) initially before randomization and at the end of the study. The control group will receive the established recommended standard physiotherapeutic treatment, including respiratory supportive therapy, chest muscle mobilization, coordination and stability training as well as walking exercise units. The training group will additionally undergo five spiroergometry- guided training sessions on ergometer per week. Three training sessions will consist of interval training; the other two sessions will consist of endurance training. Interval training hereby consists of training unit of 30 seconds at VO2 peak (maximal oxygen uptake) followed by 60 seconds below the anaerobic threshold (VT1). Endurance training units will consist of training below VT1. Criteria to stop exercise include patient exertion (Borg scale > 14), reduction in LVAD pump flow, pump speed or pump power. Both groups will perform CPET and 6 minute walk test (6 MWT) at study initiation and at study end. The training group will perform CPET including blood gas analysis every two weeks in order to adjust their individual training protocol.

ELIGIBILITY:
Inclusion Criteria:

* new implanted LVAD
* current treatment in Hospital
* hemodynamically stable patients without i.v. ionotropic Treatment
* at hand echocardiogram
* at hand spirometry
* spiroergometry including blood gas analysis.

Exclusion Criteria:

* serious psychologic/ psychiatric disorders
* breastfeeding/ pregnancy
* serious neurologic disorders
* serious comorbidities that would compromise patient compliance
* missing written informed consent
* persistent inotropic therapy
* acute or enduring infections.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Patients with a first implanted left ventricular assist device (LVAD)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in constant work rate exercise time (cwret) at 75% of patients' peak workrate. | 24 months
  Patients undergo a ramp exercise test up to maximal tolerance. A second test is performed at constant workrate which equals 75% of the achieved maximal workrate during the ramp test.

SECONDARY OUTCOMES:
Change in VO2 Peak (ml/min/kg) after training | 24 months
  A ramp test will be performed at baseline and at the end of the training program. Changes in weight adapted values (ml/min/kg) will be assessed.
Change in VE/VCO2 slope after training | 24 months
  A ramp test will be performed at baseline and at the end of the training program. Changes in the Ratio of Minute Ventilation vs. carbon dioxide Output will be assessed
Safety of the structured training program | 24 months
  All adverse and serious Events will be recorded in the training and in the Control Group. Comparison between Groups will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No